CLINICAL TRIAL: NCT01190540
Title: Cost Effectiveness of Building Capacity of Mid-level Practitioners in Sub-Saharan Africa for the Care and Prevention of HIV, Tuberculosis, Malaria and Related Infectious Diseases
Brief Title: Integrated Infectious Disease Capacity-Building Evaluation
Acronym: IDCAP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: Makerere University (Other); Accordia Global Health Foundation (Other)
Responsible Party: Principal Investigator, Marcia Weaver, Research Associate Professor, University of Washington
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 42657-EG
Record Dates: First submitted 2010-08-25; First posted 2010-08-27 (Estimated); Last update posted 2014-12-03 (Estimated); Status verified 2014-12

CONDITIONS: Capacity Building; Support for Midlevel Health Professionals; Diagnostic Training
Keywords: On site support services.; mid level health professionals.; cost effectiveness.; infectious disease.; capacity building.
MeSH Terms: conditions — Communicable Diseases | interventions — Organization and Administration

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- OSS Phase 1 (Active Comparator): Thirty-six sites will receive the On Site Support service (OSS) activities for nine to 15 months; 18 will be randomly assigned to receive the OSS in phase 1
  Interventions: Behavioral: Training and supervision; Behavioral: Integrated Management of Infectious Disease (IMID)
- OSS Phase 2 (Active Comparator): Thirty-six sites will receive the OSS activities for nine to 15 months; 18 will be randomly assigned to receive the OSS in phase 2 that will serve as a control group in phase 1 and receive OSS nine months later.
  Interventions: Behavioral: Training and Supervision; Behavioral: Integrated Management of Infectious Disease (IMID)

INTERVENTIONS:
Behavioral: Training and supervision — On-Site-Support (OSS) service training will occur monthly for a period of 9 months. This training and supervision will support the proper utilization of newly learned clinical skills.
  Arms: OSS Phase 1
Behavioral: Training and Supervision — On-Site-Support (OSS) service training will occur monthly for a period of 9 to 15 months. This training and supervision will support the proper utilization of newly learned clinical skills and continuous quality improvement of processes of care. For the control group, the OSS training will occur during phase 2, after a randomly assigned wait list control period.
  Arms: OSS Phase 2
Behavioral: Integrated Management of Infectious Disease (IMID) — The IMID is a 9-month training program that begins with a three-week course at the Infectious Diseases Institute (IDI) in Kampala Uganda. After the course participants engage in 12 weeks of distance learning followed by a one-week boost course at the IDI. Then the engage in 12 more weeks of distance learning and a final one-week boost course. This intervention is offered to two clinicians (clinical officers or registered nurses or midwives) at every OSS Phase 1 and OSS Phase 2 site.
  Arms: OSS Phase 1
Behavioral: Integrated Management of Infectious Disease (IMID) — The IMID is a 9-month training program that begins with a three-week course at the Infectious Diseases Institute (IDI) in Kampala Uganda. After the course participants engage in 12 weeks of distance learning followed by a one-week boost course at the IDI. Then the engage in 12 more weeks of distance learning and a final one-week boost course. This intervention is offered to two clinicians (clinical officers or registered nurses or midwives) at every OSS Phase 1 and OSS Phase 2 site.
  Arms: OSS Phase 2

SUMMARY:
This evaluation aim is to investigate a cost-effective way to build capacity for the care and prevention of infectious diseases among mid-level practitioners (MLP) in sub-Saharan Africa. Classroom based training continues to be the dominant form of training, despite evidence that suggests that on-site support (OSS) is more beneficial. Definitive evidence that on-site support is the most effective way to deliver the required outputs and related outcomes is still lacking. IDCAP will provide two interventions that integrate training in TB, HIV/AIDS and malaria as well as other infectious diseases, and the effects will be studied: 1) Integrated Management of Infectious Disease (IMID) training program for individual MLP, and 2) On-site support (OSS) for team of health professionals. This study employs a mixed design with pre/post and cluster randomized trial components. Interventions are at the level of the individual participant for IMID and at the level of the site (health facility) for OSS. All participants attend a 3-week course, followed by two 1-week booster courses over a six month period. After the 3-week course, a randomized arm of half the sampled facilities also received OSS every month for 9 months and bi-monthly for 6 additional months.

DETAILED DESCRIPTION:
There are four major components of the evaluation design as described below: 1) Site Assessment, 2) Competence and practice of individual MLP who participate in IDT, 3) Facility cost and performance indicators, and 4) Mortality survey. The site assessment guided the curriculum development and site selection. As shown in Figure 1, it occurred only once in Year 1. The effect of the IMID and OSS on competence of individual MLP will be evaluated with written case scenarios or vignettes. Data on case scenarios will be collected three times: a) before training, b) after the three-week course, and c) after the nine-month program that includes two, one-week booster courses and distance learning. To estimate the effect of IMID, aggregate changes in test score across all 3 time points for both arms will be analyzed jointly. To estimate the effect of OSS, differences in change in test score starting from after the three-week course to the end of the nine-month program will be compared across the 2 arms. The effects on practice of individual trainees will be evaluated with clinical assessments by mobile team faculty during five outpatients visits and five HIV clinic visits by individual MLP. Data on clinical assessments will be collected two times: a) before training, and b) after the nine-month program. Facility performance indicators will be collected on a monthly basis from each site. Sites will be randomly assigned to begin OSS in either Phase 1 or Phase 2 and the facility indicators of these two samples of sites will be compared. The principal investigators of IDCAP are actively considering collecting data on mortality among children under five, but a final decision has not been made. At the request of the acting chairperson of SOMREC, we are including information about this potential activity. Mortality surveys would be conducted before and after the OSS.

ELIGIBILITY:
Inclusion Criteria:

Facilities selected for OSS:

* The health facility had to be a HC IV or comparable facility such as a small general hospital or non-governmental organization clinic
* It had to be an active ART site or accredited ART site that is scheduled to become active by April 2009
* No past or current participation in a partnership with the U.S. Department of Defense
* Has a population of potential patients who are not prisoners
* Representation from all six administrative regions of Uganda

Exclusion Criteria:

* NA

MLP selected from the participating facilities for IMID:

Two mid-level practitioners (clinical officers, nurses, or midwives) who are actively engaged in clinical infectious-disease care will be selected for enrollment in IMID

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2008-11; Primary Completion 2012-08 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
Model of Integrated Capacity Building Program | monthly over 3 years
  The principal output of this evaluation will be a proven model of an integrated capacity-building package for the care and prevention of infectious disease in Africa. The package will include a single curriculum for MLP and a portfolio of on-site support services founded on Accordia Global Health Foundation's considerable experience in training clinicians in North America and Africa.
Competence of individual clinicians | 3 observations at pre/post IMID and final
  Competence of individual clinicians will be measured by scores on 12 written case scenarios or vignettes. Three blocks of 4 scenarios each covered different aspects of HIV/AIDS, tuberculosis, malaria, and other infectious diseases and included cases involving children, adults, and pregnant women. Each case scenario addressed 6 principal domains: emergency or danger signs, history and physical examination, laboratory testing, diagnosis or classification of patients' medical problems; initial treatment or referral plan, and evolution of the case over time.
Practice of individual clinicians | Baseline and Endline (9 months)
  Clinical assessments will be conducted by mobile team faculty who will observe individual clinicians during five outpatient visits with children under five years and five HIV clinic visits. Clinical practice will be assessed on history, physical examination, review of medical records (HIV clinic only), laboratory investigations ordered, diagnosis, treatment prescribed and patient education.
Clinical performance indicators | Monthly beginning 5 months before OSS
  54 clinical performance indicators used by the Ministry of Health, the Uganda Malaria Surveillance Program or recommended by international organizations will be used to measure performance in general areas: 1) HIV prevention, 2) HIV care, 3) Antiretroviral therapy, 4) TB/HIV care, 5) Case management of respiratory infections, 6) Case Management of Fever, and 7) Emergency Triage and Treatment.

SECONDARY OUTCOMES:
Reduce Infection, Illness, and Mortality Rates | 3 years
  The population in the areas surrounding the proposed sites will benefit directly from lower infection, illness and mortality rates. The improved ability of clinic staff to deliver quality prevention and care services will increase access to cost-effective interventions delivered according to national guidelines by 9% to 25% depending on the intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Marcia Weaver, PhD, Principal Investigator — University of Washington; Sarah Naikoba, BMBCh, MPH, Principal Investigator — Infectious Disease Institute, Makarere University
Locations (1):
- Infectious Disease Institute, Makerere University, Kampala, Uganda

REFERENCES:
- [Background] Weaver M, Krieger J, Castorina J, et. al.
- [Background] World Health Organization. Generalized Cost-Effeciveness Analysis: A Guide. Geneva: World Health Organization, 2003. Available online at: http://www.who.int/choice/en/ Accessed on April 14, 2008.
- [Background] The Uganda Bureau of Statistics (UBOS), Macro International Inc., and MEASURE Evaluation. 2008. Uganda Child Verbal Autopsy Study 2007. Calverton, Maryland, USA: UBOS, Macro International Inc., and MEASURE Evaluation.
- [Derived] Weaver MR, Crozier I, Eleku S, Makanga G, Mpanga Sebuyira L, Nyakake J, Thompson M, Willis K. Capacity-building and clinical competence in infectious disease in Uganda: a mixed-design study with pre/post and cluster-randomized trial components. PLoS One. 2012;7(12):e51319. doi: 10.1371/journal.pone.0051319. Epub 2012 Dec 14. PMID 23272097
- See also: Accordia Global Health Foundation — http://accordiafoundation.org/
- See also: Infectious Disease Institute, University of Makerere — http://idi-makerere.com/